CLINICAL TRIAL: NCT06671470
Title: Drug Interaction Study of YZJ-1139 Tablets With Ticagrelor Tablets
Brief Title: A Drug-drug Interaction Study of YZJ-1139 Tablets and Ticagrelor Tablets in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-1139-1-13
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: Single dose
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental)
  Interventions: Drug: YZJ-1139 tablets; Drug: Ticagrelor Tablets

INTERVENTIONS:
Drug: YZJ-1139 tablets — Oral dose 20 mg
Drug: Ticagrelor Tablets — Oral dose 90 mg twice daily

SUMMARY:
Primary Objective :

To evaluate the effect of ticagrelor tablets on the pharmacokinetic characteristics of YZJ-1139 in healthy subjects;

Secondary Objective:

To evaluate the safety of ticagrelor tablets in combination with YZJ-1139 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and are willing to strictly follow the clinical trial protocol to complete this trial and sign the informed consent form; 2) Male and female subjects aged 18~45 years (including cut-off value); 3) Male weight ≥ 50.0kg, female weight ≥ 45.0kg, body mass index (BMI) within the range of 19.0~26.0kg/m2 (including the cut-off value); 4) normal or abnormal physical examination, vital signs, 12-lead ECG, laboratory tests are not clinically significant; 5) Good health, those who with no respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, psychiatric system history of serious and chronic diseases; 6) Subjects (including partners) have no fertility plan, sperm/egg donation plan and voluntarily use adequate contraception from signing informed consent and within 3 months after the last dose.

Exclusion Criteria:

1. Allergies: Those with a history of two or more drug or food allergies in the past; or those who are known to be allergic to YZJ-1139 tablets and test concomitant drugs and excipients;
2. Those who have difficulty swallowing tablets, or those who have special dietary requirements and cannot accept the standard diet provided by the research center;
3. Those who cannot tolerate venipuncture, or have a history of fainting blood or needles;
4. Those who have a history or current narcolepsy, obstructive sleep apnea, complex sleep behaviors (such as sleepwalking, dream driving, etc.), severe unconscious hypoglycemia, stroke, epilepsy and other psychiatric neurological diseases (including anxiety, depression, etc.), convulsive diseases, cataplexy;
5. Those with bleeding tendency (such as recent trauma, recent surgery, coagulation dysfunction, active or recent intestinal bleeding), have a history of active pathological bleeding, intracranial hemorrhage, or other diseases that can change or increase bleeding tendency (peptic ulcer, Henoch-Schonlein purpura, lupus erythematosus, etc.);
6. Those who with abnormal clinical significance in the determination of hepatitis B surface antigen, hepatitis C virus antibody, hepatitis C virus core antigen, human immunodeficiency virus (HIV) antigen antibody combined detection, and treponema pallidum specific antibody determination;
7. Regular drinkers within 6 months prior to screening, i.e., drinking an average of more than 14 units of alcohol per week (1 unit ≈ 360mL of beer or 45mL of spirits with 40% alcohol or 150mL of wine) or > alcohol breath test results during the screening period0mg/100mL;
8. Those who have used soft drugs (such as marijuana) within 3 months before screening or taken hard drugs (such as cocaine, amphetamines, phencyclidine ) within 1 year before screening; or those with a history of substance abuse; or those who have a positive drug abuse screen at screening;
9. Those who have smoked ≥5 cigarettes per day within 3 months before screening or cannot stop using any tobacco products during the trial;
10. Those who have donated blood or lost a large amount of blood (> 400mL) within 3 months prior to screening, received blood transfusion or used blood products;
11. Those who have participated in any clinical trial and been given investigational drugs or investigational medical devices within 3 months prior to screening; or those who plan to participate in other clinical trials during the study period;
12. Those who have undergone surgical procedures within 30 days prior to screening, or who plan to undergo surgical procedures during the study;
13. Received vaccination within 30 days prior to screening, or planned vaccination during the trial;
14. Use of any drug that inhibits or induces hepatic metabolism of the drug within 28 days prior to screening (e.g.: inducers-barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; Inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines);
15. Those who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, or Chinese herbal medicines within 14 days before screening;
16. Consumption of grapefruit, pomelo, dragon fruit, mango and other fruits or related products that affect metabolic enzymes within 7 days before screening;
17. Intake of caffeine- or xanthine-rich beverages or foods (such as coffee, strong tea, chocolate, cola, etc.) within 24 hours before administration;
18. Female subjects who are lactating or have a positive pregnancy result;
19. Those who have sudden acute illness or new concomitant medication from the screening stage to before enrollment;
20. In the opinion of the investigator, the subject is not suitable for inclusion in this trial for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of YZJ-1139(Cmax) | 48 hours
  To evaluate the potential effect of multiple oral doses of ticagrelor on the single-dose PK of YZJ-1139. Maximum observed concentration (Cmax).
Pharmacokinetics of YZJ-1139 (AUC0-∞) | 48 hours
  To evaluate the potential effect of multiple oral doses of ticagrelor on the single-dose PK of YZJ-1139. Area under the concentration-time curve (AUC) from time zero to infinity.
Pharmacokinetics of YZJ-1139 (AUC0-t) | 48 hours
  To evaluate the potential effect of multiple oral doses of ticagrelor on the single-dose PK of YZJ-1139. Area under the concentration-time curve (AUC) time zero to last quantifiable concentration.

SECONDARY OUTCOMES:
Number of participants with adverse events | 13 days
  The safety and tolerability of YZJ-1139 alone and in combination with ticagrelor will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Shulan (Hangzhou) Hospital, Huangzhou, China